CLINICAL TRIAL: NCT03405870
Title: The LIPid Intensive Drug Therapy for Sepsis ¬Pilot (LIPIDS-P) Phase I/II Trial
Brief Title: LIPIDS-P Trial Phase I/II Trial
Acronym: LIPIDS-P
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201800027 - A; OCR19642 (Other: UF OnCore)
Record Dates: First submitted 2018-01-12; First posted 2018-01-23 (Actual); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-02

CONDITIONS: Sepsis, Severe; Septic Shock
Keywords: cholesterol; lipids; total parenteral nutrition
MeSH Terms: conditions — Sepsis; Shock, Septic; Hyperphagia | interventions — SMOFlipid; Parenteral Nutrition, Total

STUDY DESIGN:
Intervention Model Description: The study has a Phase I/II design. For the Phase I study, 10 patients were enrolled, and 9 completed the study. The Phase I study was designed to test the maximum tolerated dose of Smoflipid in escalating doses from 1.0 g/kg, 1.2 g/kg, 1.4 g/kg, and 1.6 g/kg. One patient withdrew from the study for social reasons. The Phase II trial was a randomized clinical trial to test the efficacy of 3 doses of study drug (1.2 g/kg, 1.4 g/kg, and 1.6 g/kg) for the primary outcome of cholesterol stabilization at 48 hours. 49 patients were enrolled and randomized. Two patients were withdrawn prior to drug. 47 patients completed the study protocol. Trial patients were randomized to receive either Smoflipid or control (no active treatment) using a Bayesian Optimal Interval Design. Thus, the Phase II arm included 24 patients in the control arm and 23 patients randomized to one of the three most efficacious doses of the study drug based on body weight, while the control group received no drug.
Who Masked: Outcomes Assessor
Masking Description: Because this is a pilot study, and because the lipid emulsion appears white and was visible to the treatment team, the study was not blinded. Data abstractors were blinded to the treatment effect. As the treatment effects are objective measurements (lipid levels, SOFA score, etc.) the likelihood of bias is low.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Phase II - 1.2 g/kg Smoflipid (Experimental): Infusion of drug (Smoflipid) will occur over a 10-16.5 hour period given once per day for the first two days of study enrollment.
  Interventions: Drug: Smoflipid
- Phase II - 1.4 g/kg Smoflipid (Experimental): Infusion of drug (Smoflipid) will occur over a 10-16.5 hour period given once per day for the first two days of study enrollment.
  Interventions: Drug: Smoflipid
- Phase II - 1.6 g/kg Smoflipid (Experimental): Infusion of drug (Smoflipid) will occur over a 10-16.5 hour period given once per day for the first two days of study enrollment.
  Interventions: Drug: Smoflipid
- Phase II - Control (No Intervention): No drug, patients will be followed as active controls
- Phase I - 1.0 g/kg Smoflipid (Experimental): Infusion of drug (Smoflipid) will occur over a 10-16.5 hour period given once per day for the first two days of study enrollment.
  Interventions: Drug: Smoflipid
- Phase I - 1.2 g/kg Smoflipid (Experimental): Infusion of drug (Smoflipid) will occur over a 10-16.5 hour period given once per day for the first two days of study enrollment.
  Interventions: Drug: Smoflipid
- Phase I - 1.4 g/kg Smoflipid (Experimental): Infusion of drug (Smoflipid) will occur over a 10-16.5 hour period given once per day for the first two days of study enrollment.
  Interventions: Drug: Smoflipid
- Phase I - 1.6 g/kg Smoflipid (Experimental): Infusion of drug (Smoflipid) will occur over a 10-16.5 hour period given once per day for the first two days of study enrollment.
  Interventions: Drug: Smoflipid

INTERVENTIONS:
Drug: Smoflipid — Administration of lipid injectable emulsion
  Other Names: Total parenteral nutrition
  Arms: Phase I - 1.0 g/kg Smoflipid; Phase I - 1.2 g/kg Smoflipid; Phase I - 1.4 g/kg Smoflipid; Phase I - 1.6 g/kg Smoflipid; Phase II - 1.2 g/kg Smoflipid; Phase II - 1.4 g/kg Smoflipid; Phase II - 1.6 g/kg Smoflipid

SUMMARY:
Briefly, this pilot clinical trial will evaluate preliminary safety and efficacy of the study drug (Smoflipid) at elevating cholesterol levels (primary outcome) in patients with sepsis and moderate organ dysfunction and will also evaluate measures of organ dysfunction, mortality, and biological activity (secondary outcomes).

DETAILED DESCRIPTION:
Sepsis is a life-threatening disease for which there are no effective treatments. It results from metabolic and immunologic derangements that lead to organ dysfunction, shock and sometimes death. Both "good" (high density lipoprotein, HDL) and "bad" (low density lipoprotein, LDL) cholesterol should be protective against sepsis by helping to clear bacterial toxins from the blood stream and by providing a fuel for endogenous corticosteroids, part of the body's protective stress-response in shock. However, for partially unknown reasons, cholesterol levels drop to critically low levels in early sepsis, leaving the body unable to protect itself against sepsis via these mechanisms. Currently, lipid emulsions are available that are FDA approved for intravenous nutrition in critically ill patients (including sepsis) and may be capable of elevating serum cholesterol levels. This Phase II randomized pilot clinical trial, proposes to assess the following in a cohort of patients with early sepsis (first 24 hours): 1) safety and tolerability of the proposed lipid injectable emulsion (Smoflipid) and any adverse effects, 2) the drugs ability to optimally elevate cholesterol at 48 hours, and 3) preliminary measures of biological activity and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. age > 18,
2. primary diagnosis of sepsis and within 24 hours of sepsis recognition and treated with institutional sepsis algorithm,
3. SOFA score ≥ 4,
4. screening total cholesterol ≤ 100 mg/dL or HDL-C + LDL-C ≤ 70 mg/dL

Exclusion Criteria:

1. total bilirubin > 2 mg/dL,
2. serum albumin < 1.5 mg/dL,
3. hypersensitivity to fish, egg, soybean, or peanut protein, or to any of the active ingredients or excipients,
4. severe hyperlipidemia or severe disorders of lipid metabolism with serum triglycerides > 400 mg/dL,
5. alternative/confounding diagnosis causing shock or critical illness (e.g., myocardial infarction or pulmonary embolus, massive hemorrhage, trauma),
6. significant traumatic brain injury (evidence of neurologic injury on CT scan and a GCS <8),
7. refractory shock (likely death within 12 hours),
8. established Do Not Resuscitate status or advanced directives restricting aggressive care or treating physician deems aggressive care unsuitable,
9. anticipated requirement for surgery that would interfere with drug infusion,
10. severe primary blood coagulation disorder,
11. acute pancreatitis accompanied by hyperlipidemia,
12. acute thromboembolic disease,
13. uncontrollable source of sepsis (e.g., irreversible disease state such as unresectable dead bowel),
14. severe immunocompromised state (e.g. subject has neutropenia receiving cytotoxic chemotherapy with absolute neutrophil count < 500/ul or expected to decline to < 500/uL within the next 3 days),
15. pregnancy or lactation
16. already receiving intravenous lipid formulations (e.g., TPN, propofol) will be excluded from the study as lipid infusion will interfere with interpretation of the study results.
17. Child Pugh Class B/C liver disease patients or liver transplant recipient
18. Patients on, or anticipated to be placed on, ECMO within 48 hours of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faheem W Guirgis, MD, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - Department of Emergency Medicine, UF Health, Gainesville, Florida
  - UF Health Emergency Medicine, Gainesville, Florida
  - UF Health Jacksonville North campus, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Augustin B, Wu D, Black LP, Bertrand A, Sulaiman D, Hopson C, Jacob V, Shavit JA, Hofmaenner DA, Labilloy G, Smith L, Cagmat E, Graim K, Datta S, Reddy ST, Guirgis FW. Multiomic molecular patterns of lipid dysregulation in a subphenotype of sepsis with higher shock incidence and mortality. Crit Care. 2024 Dec 24;28(1):431. doi: 10.1186/s13054-024-05216-3. PMID 39716214
- [Derived] Guirgis FW, Black LP, Henson M, Bertrand A, DeVos E, Ferreira J, Gao H, Wu SS, Leeuwenburgh C, Moldawer L, Moore F, Reddy ST. The Lipid Intensive Drug Therapy for Sepsis Phase II Pilot Clinical Trial. Crit Care Med. 2024 Aug 1;52(8):1183-1193. doi: 10.1097/CCM.0000000000006268. Epub 2024 Mar 15. PMID 38488429
- [Derived] Guirgis FW, Black LP, DeVos E, Henson M, Ferreira J, Miller T, Rosenthal M, Leeuwenburgh C, Kalynych C, Moldawer L, Jones L, Crandall M, Reddy ST, Gao H, Wu S, Moore F. Lipid intensive drug therapy for sepsis pilot: A Bayesian phase I clinical trial. J Am Coll Emerg Physicians Open. 2020 Nov 18;1(6):1332-1340. doi: 10.1002/emp2.12237. eCollection 2020 Dec. PMID 33392541
- [Derived] Guirgis FW, Black LP, Rosenthal MD, Henson M, Ferreira J, Leeuwenburgh C, Kalynych C, Moldawer LL, Miller T, Jones L, Crandall M, Reddy ST, Wu SS, Moore FA. LIPid Intensive Drug therapy for Sepsis Pilot (LIPIDS-P): Phase I/II clinical trial protocol of lipid emulsion therapy for stabilising cholesterol levels in sepsis and septic shock. BMJ Open. 2019 Sep 18;9(9):e029348. doi: 10.1136/bmjopen-2019-029348. PMID 31537565

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study has a Phase II design. After evaluating for DLT, 49 enrolled (2 withdrawals) with 47 patients completing the Phase II study to either Smoflipid (intervention) or control. Only Phase II data are reported here.
Groups:
- Phase II - 1.2 g/kg Smoflipid; Phase I - 1.2 g/kg Smoflipid: These patients recieved 1.2 g/kg of smoflipid.
- Phase II - 1.4 g/kg Smoflipid; Phase I - 1.4 g/kg Smoflipid: These patients recieved 1.4 g/kg of smoflipid.
- Phase II - 1.6 g/kg Smoflipid; Phase I - 1.6 g/kg Smoflipid: These patients recieved 1.6 g/kg of smoflipid.
- Phase II - Control: Active Control
- Phase I - 1.0 g/kg Smoflipid: These patients recieved 1.0 g/kg of smoflipid.
Period: Overall Study
Arm/Group | Phase II - 1.2 g/kg Smoflipid | Phase II - 1.4 g/kg Smoflipid | Phase II - 1.6 g/kg Smoflipid | Phase II - Control | Phase I - 1.0 g/kg Smoflipid | Phase I - 1.2 g/kg Smoflipid | Phase I - 1.4 g/kg Smoflipid | Phase I - 1.6 g/kg Smoflipid
Started | 11 | 4 | 10 | 24 | 2 | 2 | 3 | 3
Completed | 10 | 4 | 9 | 24 | 2 | 2 | 2 | 3
Not Completed | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: 10 patients were enrolled in the Phase I trial. One patient was withdrawn leaving nine patients for analysis. 49 patients were enrolled in the Phase II trial. Two patients were withdrawn leaving 47 patients who completed the study and were included in the analysis.
Groups:
- Phase II - 1.2 g/kg Smoflipid; Phase II - 1.4 g/kg Smoflipid; Phase II - 1.6 g/kg Smoflipid; Phase I - 1.0 g/kg Smoflipid; Phase I - 1.2 g/kg Smoflipid; Phase I - 1.4 g/kg Smoflipid; Phase I - 1.6 g/kg Smoflipid: Infusion of drug (Smoflipid) will occur over a 16.5 hour period given once per day for the first two days of study enrollment.
  Smoflipid: Administration of lipid injectable emulsion
- Phase II - Control: Patients will be followed as active controls, cholesterol levels and labs for lipid measures will be drawn.
- Total: Total of all reporting groups
Arm/Group | Phase II - 1.2 g/kg Smoflipid | Phase II - 1.4 g/kg Smoflipid | Phase II - 1.6 g/kg Smoflipid | Phase II - Control | Phase I - 1.0 g/kg Smoflipid | Phase I - 1.2 g/kg Smoflipid | Phase I - 1.4 g/kg Smoflipid | Phase I - 1.6 g/kg Smoflipid | Total
Number analyzed (Participants) | 10 | 4 | 9 | 24 | 2 | 2 | 2 | 3 | 56
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Age, y | 71 [59 to 76] | 63 [61 to 67] | 67 [48 to 77] | 68 [60 to 73] | 66 [65 to 67] | 53 [42 to 64] | 53 [44 to 63] | 59 [58 to 62] | 65 [57 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 0 | 2 | 10 | 1 | 0 | 1 | 2 | 24
  Male | 2 | 4 | 7 | 14 | 1 | 2 | 1 | 1 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 2 | 5 | 11 | 1 | 1 | 0 | 1 | 26
  White | 5 | 1 | 4 | 12 | 1 | 1 | 2 | 2 | 28
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 4 | 9 | 24 | 2 | 2 | 2 | 3 | 56

OUTCOME MEASURES:

1. Primary Outcome: Phase II - Primary Outcome - Change in Total Cholesterol (48 Hours - Enrollment)
Description: Change in total cholesterol (48 hour - enrollment value) of 0 to +5 mg/dL
Time Frame: 48 hours
Population: Phase II participants were analyzed for the primary outcome of change in total cholesterol at 48 hours (47 patients) at doses of 1.2, 1.4 and 1.6 g/kg. Phase I participants were also analyzed for this outcome, although it was not the primary outcome for this phase (which was maximum tolerated dose).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Phase II - 1.2 g/kg Smoflipid | Phase II - 1.4 g/kg Smoflipid | Phase II - 1.6 g/kg Smoflipid | Phase II - Control | Phase I - 1.0 g/kg Smoflipid | Phase I - 1.2 g/kg Smoflipid | Phase I - 1.4 g/kg Smoflipid | Phase I - 1.6 g/kg Smoflipid
Number analyzed (Participants) | 10 | 4 | 9 | 24 | 2 | 2 | 2 | 3
mg/dL | 9 (17) | -10 (29) | 4 (21) | 2 (18) | -12 (23) | 16 (1) | -9 (10) | -18 (9)

2. Primary Outcome: Phase I - Primary Outcome - Maximum Tolerated Dose/Participants Experiencing Dose Related Toxicity
Description: Using sequential dose escalation, participants received 2 doses of 1.0 to 1.6 g/kg of lipid emulsion (Smoflipid 20% lipid emulsion) within 48 hours of enrollment to test the maximum tolerated dose of study drug. The maximum tolerated dose was defined by patients exhibiting specific dose-related toxicities from administration of escalating doses of the study drug. Of 9 patients, adverse events were only considered dose-limiting toxicities if they met the predefined study protocol criteria. None of these were classified as dose limiting or serious.
Time Frame: First 48 hours
Population: Only Phase I trial patients were analyzed for this component of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II - 1.2 g/kg Smoflipid | Phase II - 1.4 g/kg Smoflipid | Phase II - 1.6 g/kg Smoflipid | Phase II - Control | Phase I - 1.0 g/kg Smoflipid | Phase I - 1.2 g/kg Smoflipid | Phase I - 1.4 g/kg Smoflipid | Phase I - 1.6 g/kg Smoflipid
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Phase I - 1.0 g/kg Smoflipid vs Phase I - 1.2 g/kg Smoflipid vs Phase I - 1.4 g/kg Smoflipid vs Phase I - 1.6 g/kg Smoflipid; Using sequential dose escalation, participants received 2 doses of 1.0 to 1.6 g/kg of lipid emulsion (Smoflipid 20% lipid emulsion) within 48 hours of enrollment to test the maximum tolerated dose of study drug. The maximum tolerated dose was defined by patients exhibiting specific dose-related toxicities from administration of escalating doses of the study drug. Of 9 patients, adverse events were only considered dose-limiting toxicities if they met the predefined study protocol criteria; Test type: Other — Determined maximum tolerated dose; Value of Maximum Tolerated Dose (g/kg) = 1.6

3. Secondary Outcome: Phase II - Secondary Outcome - Organ Dysfunction
Description: Sequential Organ Failure Assessment (SOFA) Score, this is a numerical score ranging from 0 to 24. A Higher SOFA score represents worsening organ dysfunction is correlated with higher rate of mortality. We measured the change over 48 hours.
Time Frame: 48 hours
Population: Phase I and II participants were analyzed for this secondary outcome of change in SOFA score from 0 to 48 hours.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Phase II - Control: Active control, no drug
Arm/Group | Phase II - 1.2 g/kg Smoflipid | Phase II - 1.4 g/kg Smoflipid | Phase II - 1.6 g/kg Smoflipid | Phase II - Control | Phase I - 1.0 g/kg Smoflipid | Phase I - 1.2 g/kg Smoflipid | Phase I - 1.4 g/kg Smoflipid | Phase I - 1.6 g/kg Smoflipid
Number analyzed (Participants) | 10 | 4 | 9 | 24 | 2 | 2 | 2 | 3
score on a scale | 1 [-2 to 1] | 0 [-5 to 0] | -2 [-3 to -2] | -2 [-4 to -1] | 4 [3 to 4] | -5 [-6 to -4] | -2 [-3 to 0] | 0 [-2 to 2]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from enrollment through 28 days after enrollment.
Description: Adverse events were any unfavorable and unintended sign, symptom, or disease temporally associated with the use of Smoflipid in this study. Adverse events were only considered dose-limiting toxicities if they met the predefined study protocol criteria. None of the these were classified as dose limiting or serious.
Arm/Group | Phase II - 1.2 g/kg Smoflipid | Phase II - 1.4 g/kg Smoflipid | Phase II - 1.6 g/kg Smoflipid | Phase II - Control | Phase I - 1.0 g/kg Smoflipid | Phase I - 1.2 g/kg Smoflipid | Phase I - 1.4 g/kg Smoflipid | Phase I - 1.6 g/kg Smoflipid
All-Cause Mortality (participants affected / at risk) | 1/10 | 3/4 | 0/9 | 7/24 | 1/2 | 0/2 | 0/2 | 2/3
Serious Adverse Events (participants affected / at risk) | 2/10 | 3/4 | 1/9 | 8/24 | 2/2 | 0/2 | 0/2 | 2/3
Other Adverse Events (participants affected / at risk) | 6/10 | 3/4 | 7/9 | 8/24 | 2/2 | 1/2 | 2/2 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II - 1.2 g/kg Smoflipid (N=10) | Phase II - 1.4 g/kg Smoflipid (N=4) | Phase II - 1.6 g/kg Smoflipid (N=9) | Phase II - Control (N=24) | Phase I - 1.0 g/kg Smoflipid (N=2) | Phase I - 1.2 g/kg Smoflipid (N=2) | Phase I - 1.4 g/kg Smoflipid (N=2) | Phase I - 1.6 g/kg Smoflipid (N=3)
Death (General disorders) | 1 (1) | 3 (3) | 0 (0) | 7 (7) | 1 (1) | 0 (0) | 0 (0) | 2 (2) — Unrelated, serious adverse event
Intubation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hospital Readmission (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasopressor Support (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II - 1.2 g/kg Smoflipid (N=10) | Phase II - 1.4 g/kg Smoflipid (N=4) | Phase II - 1.6 g/kg Smoflipid (N=9) | Phase II - Control (N=24) | Phase I - 1.0 g/kg Smoflipid (N=2) | Phase I - 1.2 g/kg Smoflipid (N=2) | Phase I - 1.4 g/kg Smoflipid (N=2) | Phase I - 1.6 g/kg Smoflipid (N=3)
Hyperglycemia (General disorders) | 1 (10) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Elevated triglycerides (General disorders) | 2 (2) | 0 (0) | 2 (2) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Elevated Total Bili (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (General disorders) | 2 (2) | 1 (1) | 2 (3) | 6 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased phosphorus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Line infiltration (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Elevated creatinine (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated LFT's (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated ALT (General disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated AST (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Itch (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated INR (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea and Vomiting (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
For the Phase I trial, the main limitation was the small sample of patients; however, this is not uncommon among phase I trials. The Phase II was also a small clinical trial of 47 patients, planned for 24 patients in each arm. Strict enrollment criteria limited enrollment in this study and the exclusion of patients with elevated bilirubin given the drug's hepatic metabolism and risk of complications limited the number of patients who could enroll.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/70/NCT03405870/Prot_SAP_000.pdf